CLINICAL TRIAL: NCT04343001
Title: Aspirin, Losartan and Simvastatin in Hospitalised COVID-19 Patients: a Multinational Randomised Open-label Factorial Trial
Brief Title: Coronavirus Response - Active Support for Hospitalised Covid-19 Patients
Acronym: CRASH-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Grant not obtained
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KEP-420
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: Adult Respiratory Distress Syndrome; Pneumonia; Myocardial infarction
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Pneumonia; Myocardial Infarction | interventions — Aspirin; Losartan; Simvastatin

STUDY DESIGN:
Intervention Model Description: 2 x 2 x 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Standard care (No Intervention): Usual standard of care at the study hospital
- Aspirin (Experimental): Aspirin 150mg once daily
  Interventions: Drug: Aspirin
- Losartan (Experimental): Losartan 100mg once daily. Dose may be stopped or reduced if patient is hypotensive and can be restarted anytime during the treatment period.
  Interventions: Drug: Losartan
- Simvastatin (Experimental): Simvastatin 80mg once daily
  Interventions: Drug: Simvastatin
- Aspirin and Losartan (Experimental): Aspirin 150mg once daily and Losartan 100mg once daily. Losartan dose may be stopped or reduced if patient is hypotensive and can be restarted anytime during the treatment period.
  Interventions: Drug: Aspirin; Drug: Losartan
- Aspirin and Simvastatin (Experimental): Aspirin 150mg once daily and Simvastatin 80mg once daily
  Interventions: Drug: Aspirin; Drug: Simvastatin
- Losartan and Simvastatin (Experimental): Losartan 100mg once daily and Simvastatin 80mg once daily. Losartan dose may be stopped or reduced if patient is hypotensive and can be restarted anytime during the treatment period.
  Interventions: Drug: Losartan; Drug: Simvastatin
- Aspirin, Losartan and Simvastatin (Experimental): Aspirin 150mg once daily, Losartan 100mg once daily and Simvastatin 80mg once daily. Losartan dose may be stopped or reduced if patient is hypotensive and can be restarted anytime during the treatment period.
  Interventions: Drug: Aspirin; Drug: Losartan; Drug: Simvastatin

INTERVENTIONS:
Drug: Aspirin — Aspirin 150mg
  Arms: Aspirin; Aspirin and Losartan; Aspirin and Simvastatin; Aspirin, Losartan and Simvastatin
Drug: Losartan — Losartan 100mg
  Arms: Aspirin and Losartan; Aspirin, Losartan and Simvastatin; Losartan; Losartan and Simvastatin
Drug: Simvastatin — Simvastatin 80mg
  Arms: Aspirin and Simvastatin; Aspirin, Losartan and Simvastatin; Losartan and Simvastatin; Simvastatin

SUMMARY:
The CRASH-19 trial is a multinational, open-label, factorial, randomised trial in adults hospitalised with suspected or confirmed acute COVID-19 infection.

DETAILED DESCRIPTION:
We will evaluate the effect of aspirin (150mg once daily), losartan (100mg once daily), and simvastatin (80mg once daily) in patients with COVID-19 infection.

Eligible patients will be randomly allocated to one of eight study arms (aspirin only; losartan only; simvastatin only; aspirin and losartan; aspirin and simvastatin; losartan and simvastatin; aspirin, losartan and simvastatin; standard care only). Trial treatments are given in addition to the usual standard of care at the study hospital.

Treatment will be started as soon as possible after randomisation and will continue until death, discharge or 28 days after randomisation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 40 years and older
* with suspected or confirmed acute COVID-19 infection. Acute COVID-19 infection is suspected in the presence of a fever and at least one symptom of respiratory disease e.g. cough, difficulty breathing, signs of hypoxia. The clinician may suspect COVID-19 infection if i) the patient lives in or has recently travelled to an area with COVID-19 transmission; ii) the patient had recent contact with a confirmed or probable COVID-19 case, or iii) no alternative diagnosis fully explains the clinical presentation
* requiring hospitalisation

Exclusion Criteria:

* Women known to be pregnant
* Patients hospitalised without symptoms of acute COVID-19 infection should not be recruited even if they test positive for COVID-19
* Patients already receiving mechanical ventilation
* Patients with a definite indication or contraindication for any of the trial treatments.
* Patients who are very severely frail (completely dependent and approaching end of life who typically they could not recover even from a mild illness) or terminally ill should not be recruited.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Death | up to 28 days of randomisation
  Cause of death will be described

SECONDARY OUTCOMES:
Myocardial infarction | up to 28 days of randomisation
Congestive cardiac failure | up to 28 days of randomisation
Severe cardiac arrythmia | up to 28 days of randomisation
Myocarditis | up to 28 days of randomisation
Respiratory failure including ARDS | up to 28 days of randomisation
Viral pneumonitis | up to 28 days of randomisation
Acute renal failure | up to 28 days of randomisation
Sepsis | up to 28 days of randomisation
Stroke | up to 28 days of randomisation
Gastrointestinal bleeding | up to 28 days of randomisation
Receipt of non invasive or mechanical ventilation | up to 28 days of randomisation
Ability to self care at hospital discharge | up to 28 days of randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Shakur-Still, Study Chair — London School of Hygiene and Tropical Medicine; Ian Roberts, Study Chair — London School of Hygiene and Tropical Medicine
Locations (2):
- University College Hospital, Ibadan, Oyo State, Nigeria
- Shifa Tameer-e-Millat University, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
As many sites will contribute to this trial, individual sites cannot restrict the publication of the manuscript relating to the outcomes of this trial. All anonymised data from this trial will be made freely available on our data sharing site: http://freebird.lshtm.ac.uk.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 6 months or sooner of publication
Access Criteria: Log-in required for the sole purpose to monitor data download.
URL: http://freebird.lshtm.ac.uk